CLINICAL TRIAL: NCT01255384
Title: Possible Epigenetic Changes in Offspring of Women With Pregestational and Gestational Diabetes: Molecular Studies of the Placenta and Cord Blood and Possible Correlation to Postnatal Development.
Brief Title: Possible Epigenetic Changes in Offspring of Women With Pregestational and Gestational Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Asher Ornoy, Laboratory of Teratology, Israel Canada Institute of Medical Research, Hebrew University Hadassah Medical School, Jerusalem, Israel.
Other Study IDs: EPI-DIABETES-HMO-CTIL
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Gestational Diabetes; Pregestational Diabetes; IDM (Infant of Diabetic Mothers); Neurodevelopmental Outcome; Epigenetic Changes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placental biopsy cord bloos Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non Diabetic-Controls: Pregnant women with uncomplicated pregnancy will be followed, their offsprings will be evaluated and followed for 5 years
- Diabetic Pregnancy: Pregnant women followed in the high risk clinic because of diabetes will be followed and their offspring's will be evaluated and followed for 5 years

SUMMARY:
Pregestational diabetes (PGD) during pregnancy may be associated with an increased rate of spontaneous abortions, intrauterine death and congenital anomalies among the offspring. Although the prevalence of congenital anomalies among the offspring of diabetic mothers is reduced as a result of the improvement of the glycemic control in the early pregnancy, the rate of congenital anomalies is increased and there seems to be an increased rate of neurodevelopmental disorders including some fine and gross motor deficits as well as increased rate of inattention and/or hyperactivity. In gestational diabetes, that develops in the second half of pregnancy (past the period of major organogenesis), there seems to be no increase in the rate of major congenital anomalies but there are some developmental disorders in the offspring.

The exposure of the developing embryo and fetus to diabetic environment (i.e. hyperglycemia, hyperketonemia ext), is known to cause increased oxidative stress and significant changes in gene expression as observed in several experimental diabetic models. We hypothesize that diabetic environment may also cause long lasting epigenetic changes. It is therefore our purpose to evaluate these possible epigenetic changes and correlate their presence with the degree and time of onset of diabetes, (i.e. whether from the beginning as in PGD or in the second half of pregnancy as in GD), the degree of oxidative stress and with the neurodevelopmental outcome of the offspring. Diabetic pregnancies will be compared to a similar number of normal pregnancies in all parameters studied.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to women suffering from pre-gestational or gestational diabetes.

Exclusion Criteria:

* Non Jewish population
* Triplets and up
* Premature infants under 32 weeks
* Infants suffering from major congenital anomalies
* Infants with chromosomal aberrations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants of diabetic mothers. The follow-up will start at the high risk pregnancy clinic. The obstetrician will follow women with pre-gestational and gestational diabetes. The neonates will be evaluated and followed for epigenetic changes and neurodevelopmental outcome
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Asher Ornoi, MD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel